CLINICAL TRIAL: NCT05793112
Title: Restoring Gut Health With INF108F in Infants With Food Protein Induced Allergic Proctocolitis
Brief Title: INF108F in Infants With Food Protein Induced Proctocolitis
Acronym: RESTORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Qian Yuan, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022P002752
Record Dates: First submitted 2023-03-17; First posted 2023-03-31 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-11

CONDITIONS: Infant Development; Gut Microbiome; Food Protein Induced Allergic Proctocolitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- INF108F (Experimental): INF108F
  Interventions: Drug: INF108F probiotic
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INF108F probiotic — Oral suspension
  Arms: INF108F
Drug: Placebo — Oral suspension
  Arms: Placebo

SUMMARY:
Single-center, randomized, double-blind, placebo-controlled trail evaluating INF108F in breastfed infants with FPIAP

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled trial with two arms evaluating IBF108F in breastfed infants with FPIAP. Assessments will be conducted over a 4-week study period with assessment of blood in stool, infant stooling, sleep, feeding, and growth. Safety will be evaluated through collection adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Infants, male or female, of all ethnic/racial groups, with a gestational period of 37 to 42 weeks
* Infants aged 1 - 90 days old with a documented FPIAP with either gross blood or microscopic blood in without other possible causes
* Infants must be exclusively breastfed or at least half of oral intake is from breast feeding or from expressed breast milk
* A willing parent or legal guardian will sign the consent form either electronically or with a wet ink signature

Exclusion Criteria:

* Infants born earlier than 37 weeks of gestation
* Infants who are exclusively formula-fed or less than half of oral intake is from breastfeeding or from expressed breast milk at the time of enrollment
* Infants born with medical complications (i.e., neurological, cerebral palsy, confirmed food allergies)
* Diagnosis of other severe or complicating medical problems, including autoimmune or chronic immune inflammatory conditions, gastrointestinal inflammatory conditions, or renal insufficiency
* History of abdominal surgery or congenital abnormalities of the GI track, the cardiovascular system, the pulmonary system or the renal system
* Antibiotic use (oral or systemic) within 7 days prior to enrollment
* Mother's intent to feed non-study probiotics or solid food to their infant at any time during the study
* Mothers with substance use disorder (SUD) or on Nicotine replacement therapy (NRT)
* Infants who have consumed any B. infantis-containing probiotics since birth

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Newton Wellesley Hospital, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Breastfed infants with FPIAP, w/ either grossly visible bloody stool or microscopic bloody stools, excl. other causes, will be recruited at PNW or MGH Pediatric GI clinic. They will be provided basic information about the study. We will ask potential participants to provide basic contact information and answer some study-specific questions as a pre-qualifier. Individuals who are interested to learn more will receive more details about the study, the informed consent, and study team contacts.
Period: Overall Study
Arm/Group | INF108F | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INF108F | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Weight at birth [Mean (Standard Deviation); unit: kilograms (kg)] | 3.18 (0.527) | 3.56 (0.417) | 3.37 (0.51)
Birth Mode [Count of Participants; unit: Participants]
  Vaginal | 8 | 6 | 14
  C-section | 2 | 4 | 6
Singleton delivery [Count of Participants; unit: Participants] | 10 | 10 | 20
Delivered in a Hospital [Count of Participants; unit: Participants] | 10 | 10 | 20
Maternal antibiotic exposure during labor/delivery [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 6
  No | 6 | 6 | 12
  Unknown | 1 | 1 | 2
Highest education of either parent in home is Bachelor's or Advanced degree [Count of Participants; unit: Participants] | 10 | 10 | 20
Baby ever consumed infant formula [Count of Participants; unit: Participants]
  Yes | 5 | 5 | 10
  No | 5 | 5 | 10
Baby ever consumed infant probiotics [Count of Participants; unit: Participants]
  Yes | 1 | 4 | 5
  No | 9 | 6 | 15
Baby ever consumed solid food [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 10 | 10 | 20
Baby ever consumed iron supplements [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 10 | 10 | 20
Mother ever consumed medication to treat acid reflux of GERD [Count of Participants; unit: Participants]
  Yes | 7 | 6 | 13
  No | 3 | 4 | 7
Acid reflux medication taken after baby was born [Count of Participants; unit: Participants] | 2 | 4 | 6
Type of Acid Reflux medication consumed [Count of Participants; unit: Participants]
  Famotidine | 1 | 1 | 2
  Mylanta | 0 | 1 | 1
  None | 9 | 8 | 17
Mother ever had any type of allergy [Count of Participants; unit: Participants]
  Yes | 1 | 4 | 5
  No | 9 | 6 | 15
Type of allergy (mother) [Count of Participants; unit: Participants]
  Asthma | 0 | 0 | 0
  Allergic rhinitis | 1 | 1 | 2
  Eczema | 1 | 3 | 4
  Food allergy | 0 | 1 | 1
  None | 8 | 5 | 13
Father ever had any type of allergy [Count of Participants; unit: Participants]
  Yes | 5 | 3 | 8
  No | 5 | 7 | 12
Type of allergy (father) [Count of Participants; unit: Participants]
  Asthma | 2 | 0 | 2
  Allergic rhinitis | 2 | 2 | 4
  Eczema | 3 | 1 | 4
  Food allergy | 3 | 1 | 4
  None | 0 | 6 | 6
Age, Customized [Mean (Standard Deviation); unit: Weeks]
  Age at Enrollment in weeks | 9.2 (3.29) | 9.4 (2.72) | 9.3 (3.02)
  Age at First Physical Exam in weeks | 9.1 (3.38) | 9.4 (2.27) | 9.25 (2.88)
  Gestational Age at Birth in weeks | 39.55 (0.997) | 39.55 (0.923) | 39.55 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Changes to Gut Microbiome Composition
Description: Absolute change from baseline in relative abundance of B. infantis INF108F to Study Day 28 via metagenomics results in mITT population. Unit measured: The absolute change from baseline in the percentage of sequenced reads assigned to B. infantis INF108F (calculated as value at Day 28 - value at baseline).
Time Frame: Baseline to Day 28
Population: There will be two analysis populations defined for this study. Analysis of the primary, key secondary, and other secondary endpoints will be completed on the modified Intent-to-Treat (mITT) population. All safety-related tabulations will be based upon the Safety population. The mITT population will include all infants who are randomized and receive at least one supplementation of the intervention. Infants will be analyzed according to the group to which they are randomized.
Measure: Mean (Standard Deviation); unit: Change in %B.infantis reads (Day 28-BL)
Arm/Group | INF108F | Placebo
Number analyzed (Participants) | 9 | 8
Change in %B.infantis reads (Day 28-BL) | 42.816 (53.236) | -12.413 (35.104)
Statistical Analysis 1: Comparison: INF108F vs Placebo; Test type: Superiority; p = 0.154, Wilcoxon range sum test; Median Difference (Final Values) = 57.57

2. Secondary Outcome: Changes to Clinical Symptoms of FPIAP
Description: We will collect information using questionnaires about infants' gastroesophageal reflux disease symptoms, feeding, sleep and stool frequency and consistency.
  The severity of infant GER will be quantified using the Infant Gastroesophageal Reflux Questionnaire (I-GERQ), with numeric scores. The minimum score is 0 and the maximum score is 25; scores >7 provide 74% specificity and 94% sensitivity for diagnosing GERD. Higher I-GERQ scores/values are indicative of worse outcomes, worse reflux symptoms for the infant.
  The secondary outcome was reported as the absolute change from baseline in I-GERQ score; therefore, a higher value would be positive as the score is reduced significantly from baseline, which means reflux symptoms were improved.
  The sleep will be captured using Infant Sleep Questionnaire, with 0-10 scales, 0 means worst sleep and 10 means excellent sleep for quantify the quality of infant's night sleep.
Time Frame: Baseline to day 28
Population: Analysis of the key secondary endpoints will be completed based on the modified Intent-to-Treat (mITT) population. The mITT population will include all infants who are randomized and receive at least one supplementation. Infants will be analyzed according to the group to which they are randomized.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | INF108F | Placebo
Number analyzed (Participants) | 10 | 10
Scores on a scale | -5.5 [-14 to 3] | 0.0 [-3 to 1]
Statistical Analysis 1: Comparison: INF108F vs Placebo; Test type: Superiority; p = 0.073, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -5

3. Secondary Outcome: Percentage of Infants With no Gross/Visible Blood in Stool on Study Day 14 Via the Daily Log
Description: Analysis of the key secondary endpoints will be completed based on the modified Intent-to-Treat (mITT) population. The mITT population will include all infants who are randomized and receive at least one supplementation. Infants will be analyzed according to the group to which they are randomized.
Time Frame: Enrollment to Study Day 14
Population: Percentage of infants with no gross/visible blood in stool on Study Day 14 via the daily log
Measure: Count of Participants; unit: Participants
Arm/Group | INF108F | Placebo
Number analyzed (Participants) | 10 | 10
Participants
  Gross/visible blood in stool on Day 14 | 0 | 2
  No gross/visible blood in stool on Day 14 | 10 | 8
Statistical Analysis 1: Comparison: INF108F vs Placebo; Test type: Superiority; p = 0.471, Fisher Exact; Mean Difference (Final Values) = -2

4. Secondary Outcome: Percentage of Infants Within Each Category of 'Do You Consider Your Baby's Sleep a Problem?' (Not a Problem at All, a Very Small Problem, a Small Problem, a Moderate Problem, a Serious Problem) at Baseline and Study Days 7, 14, and 28 Via the Weekly Log
Description: as for outcome 3
Time Frame: Baseline, Study Day 7, Study Day 14, Study Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | INF108F | Placebo
Number analyzed (Participants) | 10 | 10
Participants
  Day 0 (Baseline): Not a problem at all | 2 | 5
  Day 0 (Baseline): A very small problem | 1 | 3
  Day 0 (Baseline): A small problem | 4 | 1
  Day 0 (Baseline): A moderate problem | 3 | 1
  Day 0 (Baseline): A serious problem | 0 | 0
  Day 0 (Baseline): Missing | 0 | 0
  Day 7: Not a problem at all | 1 | 6
  Day 7: A very small problem | 7 | 3
  Day 7: A small problem | 2 | 0
  Day 7: A moderate problem | 0 | 1
  Day 7: A serious problem | 0 | 0
  Day 7: Missing | 0 | 0
  Day 14: Not a problem at all | 2 | 6
  Day 14: A very small problem | 3 | 2
  Day 14: A small problem | 5 | 1
  Day 14: A moderate problem | 0 | 1
  Day 14: A serious problem | 0 | 0
  Day 14: Missing | 0 | 0
  Day 21: Not a problem at all | 2 | 6
  Day 21: A very small problem | 4 | 3
  Day 21: A small problem | 1 | 0
  Day 21: A moderate problem | 2 | 1
  Day 21: A serious problem | 0 | 0
  Day 21: Missing | 1 | 0
  Day 28: Not a problem at all | 3 | 6
  Day 28: A very small problem | 3 | 2
  Day 28: A small problem | 2 | 0
  Day 28: A moderate problem | 2 | 2
  Day 28: A serious problem | 0 | 0
  Day 28: Missing | 0 | 0
Statistical Analysis 1: Comparison: INF108F vs Placebo; Day 0 (Baseline); Test type: Superiority; p = 0.057, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: INF108F vs Placebo; Day 7; Test type: Superiority; p = 0.169, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: INF108F vs Placebo; Day 14; Test type: Superiority; p = 0.168, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: INF108F vs Placebo; Day 21; Test type: Superiority; p = 0.139, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: INF108F vs Placebo; Day 28; Test type: Superiority; p = 0.348, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: From baseline to final follow-up study visit, an average of 30 days
Arm/Group | INF108F | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INF108F (N=10) | Placebo (N=10)
Failure to thrive (Metabolism and nutrition disorders) | 2 (3) | 4 (4) — Mild, dose not changed, no treatment
Colicky (Gastrointestinal disorders) | 2 (4) | 2 (5) — Mild, dose not changed, treatment with conmed
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild, dose not changed, no treatment
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild, dose not changed, no treatment
Gas (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild, dose not changed, no treatment
Mild eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild, dose not changed, no treatment
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) — Mild, dose not changed, no treatment

LIMITATIONS AND CAVEATS:
This study was a pilot study with a very limited sample size (n=20).

Not all participants were per protocol of the study with the INF108 population having two participants (20%) considered not per protocol and the placebo having one participant (10%) not per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05793112/Prot_SAP_000.pdf